CLINICAL TRIAL: NCT05394597
Title: Field Evaluation of Two Topically Applied Insect Repellent Products Containing IR3535 Against Mosquitos in Louisiana
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Kristen Healy, Associate Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4370
Record Dates: First submitted 2021-06-14; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Bites and Stings
Keywords: mosquito
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Intervention Model Description: Treatment versus control. 13 with repellent and 2 without, for 15 subjects. Median Complete Protection Time for each repellent product tested against mosquitos for prevention of biting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Receives a dose of repellent on the lower portion of the leg that is exposed
  Interventions: Other: Repellent lotion; Other: Repellent Wipe
- Control group (No Intervention): Does not receive a dose of repellent, but subject to similar exposure period

INTERVENTIONS:
Other: Repellent lotion — lotion of the repellent active ingredient IR3535
  Other Names: IR3535 Repellent in lotion format
  Arms: Treatment group
Other: Repellent Wipe — wipe of the repellent active ingredient IR3535
  Other Names: IR3535 Repellent in wipe format
  Arms: Treatment group

SUMMARY:
To determine the efficacy and duration of protection of two topically applied insect repellent products at preventing landing by mosquitos. The study will follow the EPA Product Performance Test Guidelines1. It is intended to test the products against natural populations of mosquito species of public health importance within the genera Aedes, Anopheles, and Culex, and to replace data from one site previously tested in Florida with data from a site in Louisiana with adequate landing pressure from target mosquito species of public health relevance.

DETAILED DESCRIPTION:
A single-site field setting study using healthy volunteers to test two insect repellent product formulations (lotion, and wipe) against mosquitos.

Subjects will have repellent applied to one lower limb at a standardised dose rate to account for skin area. They will then expose this area only in a field site where mosquitos are recorded landing at a rate of 5 mosquitos per 5 minute or higher. The exposure period will last five minutes and all mosquitos landing on the exposed skin will be collected using an aspirator. 5 minute exposure periods will be repeated every half hour for 14 hours for the lotion and 13 hours for the wipe, or until median CPT can be established by more than half of subjects reaching treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give fully informed consent;
* Male or female;
* Aged 18 to 55 years;
* Consider themselves to be in good general health, and specifically:

  * Not aware of having any cardiovascular or respiratory disorder (whether active or inactive)
  * No previous anaphylaxis
  * Not aware of having a compromised immune system
* Non-smokers or willing to refrain for 24 hours prior to and during each test;
* Willing to undergo a mosquito attraction test (putting an arm into a cage of mosquitos)
* Able to speak and understand English
* Able to stand outside for periods of at least 5 minutes at a time
* Able to understand and comply with the study procedures, including:

  * Willing to complete mosquito landing/aspirating training
  * Able to withstand exposing the lower leg to mosquitos for periods of at least 5 minutes at a time
  * Able to operate an aspirator

Exclusion Criteria:

* Participated in any other intervention study in the previous 3 months
* Participated in a biting insect test as part of the current study in the previous 72 hours
* Employees, managers, and spouses of employees of the LSU and of the study Sponsor (LivFul, Inc.)
* Students of the Study Director or any other LSU faculty/researchers involved in the study
* Individuals suspected or known to be sensitive or allergic to, or phobic of, mosquito bites
* Women who are pregnant, nursing or intending to become pregnant during the course of the study
* Individuals with localized skin disorders or problems affecting the legs (such as eczema, psoriasis, or atopic dermatitis) or open cuts or scrapes
* Individuals with known or suspected allergy or sensitivity to the test product or any of its ingredients, or any insect repellent products
* Individuals who are not attractive to mosquitos during mosquito attractiveness test
* Individuals who have signs or symptoms related to COVID-19, have tested positive for COVID-19 within the last 15 days, or have had contact (within 6 feet for a total of 15 minutes or more) with someone who has tested positive for COVID-19 in the last 14 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Median Complete Protection Time | 14 hours
  the time for each repellent product tested that shows efficacy against mosquito bites

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Healy, PhD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- Louisiana State University, Department of Entomology, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT05394597/Prot_000.pdf
  • Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT05394597/ICF_001.pdf